CLINICAL TRIAL: NCT05570942
Title: The Effectiveness of Oral Lactobacillus Rhamnosus TCELL-1 Upon Colorectal Cancer
Brief Title: Oral Lactobacillus Rhamnosus TCELL-1 and Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 202109062RIPD
Record Dates: First submitted 2021-12-24; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2021-12

CONDITIONS: Staged III Colorectal Cancer Receiving Adjuvant Chemotherapy

STUDY DESIGN:
Intervention Model Description: Arm 1: probiotics group; arm 2: control group (no probiotics; placebo)
Who Masked: Participant, Investigator
Masking Description: The patient were given bottle of placebo with same appearance of bottle of probiotics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Active Comparator): The patients with staged III colorectal cancer receiving adjuvant chemotherapy who will be given probiotics.
  Interventions: Dietary Supplement: Oral Lactobacillus rhamnosus TCELL-1
- Control group (Placebo Comparator): The patients with staged III colorectal cancer receiving adjuvant chemotherapy who will be given placebo.
  Interventions: Dietary Supplement: Oral Lactobacillus rhamnosus TCELL-1

INTERVENTIONS:
Dietary Supplement: Oral Lactobacillus rhamnosus TCELL-1 — A kind of probiotics which was isolated from the intestinal mucosa of health Taiwanese people

SUMMARY:
Emerging evidences have shown that gut microbiota have played roles in the modulation of chemotherapy agents for cancer patients receiving chemotherapy. Probiotics are gut microbiota beneficial to human body. However, little was known about the role of probiotics for cancer patients receiving chemotherapy. Lactobacillus rhamnosus TCELL-1 is a kind of probiotics which were isolated from the gut mucosa of healthy Taiwanese. The aim of the study was to evaluate the effect of Lactobacillus rhamnosus TCELL-1 upon staged III colorectal cancer patients receiving adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged older than 20 years (inclusive) of either gender
2. Expressed interest and ability to fulfill the study requirements.
3. Be in general good health as determined by the first evaluation within 30 days of the first dose of Lactobacillus Rhamnosus TCELL-1
4. Able to ingest the study drug (Lactobacillus Rhamnosus TCELL-1) dissolved in a small amount of cow's milk or soy milk orally (no feeding tube).
5. Willing to prevent pregnancy - Women must agree not to become pregnant or breastfeed from the time of study enrollment until at least 3 months after the last dose of study drug. If a woman is sexually active and has no history of hysterectomy or tubal ligation, she must agree to practice an acceptable method of birth control, such as hormonal or barrier birth control. A woman is eligible if she is monogamous with a vasectomized male. Sexually active male volunteers without vasectomy must agree to use a barrier method of contraception for 3 months after the last dose of study drug.
6. Willing to comply with protocol and report on compliance and side effects during study period.
7. Informed consent obtained and signed prior to screening.

Exclusion Criteria:

1. Women who are pregnant or breast-feeding or with child-bearing potential but unable or unwilling to practice a highly effective means of contraception
2. With uncontrolled infection or serious infection within the past 4 weeks
3. Patients who took antibiotics for some reasons within the past 4 weeks
4. Patients who must eat probiotics product for some reasons
5. Active substance abuse, including alcohol, which, in the opinion of the investigator, risks impairing the ability of the patient to comply with the protocol
6. History of allergy to any substance of investigational products
7. With known human immunodeficiency virus (HIV) infection
8. Judged to be not applicable to this study by investigator such as difficulty of follow-up observation
9. With any other serious diseases/medical history considered by the investigator not in the condition to enter the trial
10. Having participated other investigational study within 4 weeks of entering this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in quality of life assessed by (WHOQOL)-BREF Taiwan version | 1 year
  THE WORLD HEALTH ORGANIZATION QUALITY OF LIFE (WHOQOL)-BREF Taiwan version
Changes in quality of life assessed by EORTC QLQ-CR30 | 1 year
  EORTC QLQ-CR30
Chinese version of EORTC quality of life questionnaire(QLQ)-C30 | 1 year
The Functional Assessment of Cancer Therapy (FACT)-G version 4 | 1 year
Changes in FACT-F version 4 at each post-treatment visit compared to baseline | 1 year
Changes of irritable bowel symptoms | 1 year
  The irritable bowel symptoms will be evaluated with the Rome IV criteria of irritable bowel disease

SECONDARY OUTCOMES:
Change of fecal microbiota features | 1 year
  Fecal microbiota composition
Change of fecal metabolites | 1 year
  Fecal metabolites such as acetic acid, propionic acid, butyric acid, isobutyric acid, valeric acid and isovaleric acid
Incidence of adverse events | 1 year
  The adverse events of the probiotics
The change of body weight | 1 year
  Changes of body weight from baseline to post-treatment visits
Change of serum cytokines | 1 year
  Interleukin (IL)-1, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12, IL-13, IL-15, IL-17, interferon (IFN)-γ, tumor necrotic factor (TNF)-α3
The presence of bacteremia | 1 year
  The presence of probiotics-related bacteremia

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- Yu-Tso LIAO, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No